CLINICAL TRIAL: NCT06766370
Title: The Application of Multimodal Ultrasound Imaging in Carpal Tunnel Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dr. weijing zhang, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2024-796-01
Record Dates: First submitted 2024-12-22; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound-guided nerve hydrodissection treatment — Under ultrasound guidance, a mixed solution of corticosteroids and local anesthetics is injected around the nerve, followed by release of the transverse carpal ligament.

SUMMARY:
The aim of this study is to explore the application value of multimodal ultrasound parameters in the diagnosis and treatment follow-up of Carpal Tunnel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years;
2. Presence of sensory abnormalities and motor dysfunction in the median nerve distribution area;
3. Positive Tinel's sign or Phalen's test;
4. Neurophysiological examination consistent with mild to moderate Carpal Tunnel Syndrome.-

Exclusion Criteria:

1. Severe Carpal Tunnel Syndrome;
2. Concurrent rheumatic, metabolic, systemic, or other systemic diseases;
3. Concurrent cervical spondylosis or other peripheral neuropathies;
4. Wrist joint trauma, surgery, space-occupying lesions, or nerve itself with space-occupying lesions;
5. Concurrent malignant tumors or severe cardiopulmonary diseases;
6. History of previous wrist surgery or injections;
7. Pregnancy;
8. Allergy to corticosteroids or local anesthetics.-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study primarily utilizes ultrasound multimodal imaging to observe the changes in multiple parameter indicators before and after the treatment of nerve hydrodissection combined with transverse carpal ligament release in patients clinically diagnosed with mild to moderate Carpal Tunnel Syndrome.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire ，BCTQ | 1,3,6,12 months
  The Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome. The Symptom Severity Scale (SSS) with 11 questions is scored on a Likert scale of 1-5 and the Functional Status Scale (FSS) with 8 questions is scored from 1-5 with 1 as no difficulty and 5 as difficult.The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
the patient's sensory nerve conduction velocity (SNCV) | 3,6,12months
  SNCV in m/s
the patient's distal motor latency (DML). | 3,6,12months
  DML in ms

IPD SHARING:
Plan to Share IPD: No